CLINICAL TRIAL: NCT01727908
Title: Screening for Familial Gastric Cancer in First Degree Relatives
Acronym: FamGaCan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: guideline developed
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Protocol ID 2012/270
Record Dates: First submitted 2012-11-08; First posted 2012-11-16 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2017-04

CONDITIONS: Malignant Neoplasm of Stomach; Carcinoma, Diffuse Type; Intestinal Type Adenocarcinoma of Stomach; Relative (Related Person)
Keywords: Familial Gastric Cancer Screening
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopy without staining of the mucosa (No Intervention)
- Endoscopy with staining of the mucosa. (Experimental)
  Interventions: Other: Endoscopy with staining of the mucosa

INTERVENTIONS:
Other: Endoscopy with staining of the mucosa — Staining of the gastric mucosa with acetic acid and Indigocarmine
  Arms: Endoscopy with staining of the mucosa.

SUMMARY:
The purpose of this study is to determine whether staining of the gastric mucosa increases the number of detected (pre)malignant foci of intestinal and diffuse type gastric cancer, in first degree relatives of individuals with familial gastric cancer.

DETAILED DESCRIPTION:
Rationale:

Familial gastric cancer (FGC) concerns about 10% of all gastric cancers. It has an impressive impact on both emotional and physical wellbeing of first degree relatives of patients with (early) onset of gastric cancer. FGC can in 1-3% be attributed to one single hereditary syndrome, the hereditary diffuse gastric cancer (HDGC). HDGC is associated with a CDH1 mutation in about 40 % of the cases. In case there is no CDH1 mutation, referred to as familiar diffuse gastric cancer (FDGC), it remains uncertain how to guide and/or screen family members. The same applies for the rare familial intestinal type gastric cancer (FIGC).

Aim:

In this study we want to determine the value of endoscopic screening in members of families with FGC, both FDGC and FIGC. Also, we will analyze the associations of life style factors, including dietary habits with the development of FDGC, to be able to built preventive strategies. Finally, we want to assess the psychological impact of our screening protocol.

Objective:

Primary, to determine whether staining of the gastric mucosa increases the number of detected (pre)malignant foci of diffuse type gastric cancer, in individuals from families with FDGC as well as dysplastic, adenomatous and early intestinal cancers in individuals from families with FIGC. Secondary: A To determine the optimal pathological work-up the detection rate of (pre-)malignancy. B To determine clinical and life style factors that are associated with the two types of FGC. C To determine the psychosocial impact of the screening protocol in this population. D To develop a strategy for screening individuals from FGC families and creative advise for preventive measures.

Study design:

A randomized controlled trial included in a prospective cohort analysis.

Study population:

All (first degree) relatives , from 18 years and older from patients who fulfill the criteria for a FGC. These are; 1] all first degree relatives of an individual with diffuse gastric cancer, without proven CDH1 mutation, or members from families with 2] 2 or more individuals with gastric carcinoma, at least one < 50 yrs, or 3] 3 or more individuals with gastric carcinoma, any age, any type, or 4] 1 individual with any type gastric carcinoma < 40 yrs.

ELIGIBILITY:
Inclusion Criteria:

* adult (≥ 18 yrs), female and male relatives
* fully legal competent (to simplify the common consent agreement for blood withdrawal, DNA analysis and serial endoscopies.)
* individuals that signed the common consent agreement
* first degree relative of an individual with diffuse gastric cancer from a FDGC-family, without proven mutation,

  * OR: 2 or more individuals with gastric carcinoma, at least one < 50 yrs
  * OR: 3 or more individuals with (diffuse/intestinal/other type) gastric carcinoma, any age
  * OR 1 individual with any type gastric carcinoma < 40 yrs

Exclusion Criteria:

* immature individuals
* actual gastric ulcer or gastric bleeding
* previous diagnosis of gastric cancer
* hypersensitivity to Indigocarmine
* individuals with co-morbidity which might increase the sedation and/or endoscopy risk: COPD Gold III/IV Cardiac failure Increased bleeding tendency or use of medication which increases bleeding tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The percentage of increasement of endoscopic detection of (pre)malignant for gastric cancer by staining of the gastric mucosa. | all patients will have a follow up of five years, during which four endoscopies will be performed

SECONDARY OUTCOMES:
To determine the optimal pathological work-up the detection rate of (pre-)malignancy, measured by the number of (pre) malignant foci found by the pathologist with different coloring and immunohistochemic techniques. | all patients will have a follow up of five years, during which four endoscopies with biopsy sampling will be performed
To determine the association of clinical and life style factors with the two type of Familial Gastric Cancer, partly assessed from the patients'clinical files (eg BMI), partly by assessment of possible risk factors in blood (eg Helicobacter Pylori). | after three years of follow up these data will be assessed
To determine the psychosocial impact of the screening protocol in this population, measured as the amount of stress and anxiety by use of the Hospital Anxiety and Distress Scale and the amount of cancer-worry by use of the Cancer Worry Scale. | during the follow up period of five years, each patient will receive questionaires at six time points. Assessment of these data will be performed after finishing the follow-up of the last patient, about six years after the start of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Bisseling, M.D.Ph.D., Principal Investigator — Department of Gastroenterology and Hepatology, Radboud University Nijmegen Medical Centre; Fokko M Nagengast, M.D.Ph.D., Principal Investigator — Department of Gastroenterology and Hepatology
Locations (1):
- Department of Gastroenterology and Hepatology, Radboud University Nijmegen Medical Centre, Nijmegen, PO BOX 9101, Netherlands